CLINICAL TRIAL: NCT04705363
Title: A Sociolinguistic-enabled Web Application to Develop Precision Health Intervention for African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IRB202001790-N; UL1TR001427 (NIH)
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A 4-arm randomized experimental message design.
Who Masked: Participant, Investigator
Masking Description: Participants will be blind to condition. Investigators will be blind to which participants will be assigned to which interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Text-only (Active Comparator): A virtual health assistant that will consist of photos of the computer-generated doctor with text that will guide participants through the interaction. No voice will accompany the photos or text.
  Interventions: Behavioral: Text-only
- High Dialectal (Experimental): A virtual health assistant that will consist of an interactive computer-generated doctor with voice that used high dialectal variation that will guide participants through the interaction.
  Interventions: Behavioral: High Dialectal
- Low Dialectal (Experimental): A virtual health assistant that will consist of an interactive computer-generated doctor with voice that used low dialectal variation that will guide participants through the interaction.
  Interventions: Behavioral: Low Dialectal
- Non-Dialectal (Experimental): A virtual health assistant that will consist of an interactive computer-generated doctor with voice that used no dialectal variation that will guide participants through the interaction.
  Interventions: Behavioral: Non-Dialectal

INTERVENTIONS:
Behavioral: High Dialectal — A virtual health assistant that will consist of an interactive computer-generated doctor with voice that used high dialectal variation that will guide participants through the interaction.
  Arms: High Dialectal
Behavioral: Low Dialectal — A virtual health assistant that will consist of an interactive computer-generated doctor with voice that used low dialectal variation that will guide participants through the interaction.
  Arms: Low Dialectal
Behavioral: Non-Dialectal — A virtual health assistant that will consist of an interactive computer-generated doctor with voice that used no dialectal variation that will guide participants through the interaction.
  Arms: Non-Dialectal
Behavioral: Text-only — A virtual health assistant that will consist of photos of the computer-generated doctor with text that will guide participants through the interaction. No voice will accompany the photos or text.
  Arms: Text-only

SUMMARY:
This pilot study will explore the preliminary efficacy of a colorectal cancer (CRC) screening intervention delivered by Virtual Human Agents (VHAs). Seven hundred fifty participants aged 45 to 75 will be recruited through Qualtrics panels. The study examines how different levels of dialectal linguistic features willingness to be screened for colorectal cancer. Participants will be randomly assigned to interact with one of four VHA conditions: a VHA using non-dialectal linguistic features, a VHA with a low level of dialectal linguistic features integrated, a VHA with a high level of dialectal linguistic features integrated, or a text-only control condition. Following the interaction, participants will complete survey measures to assess perceived willingness to be screened.

DETAILED DESCRIPTION:
African Americans experience significant health inequities, including higher morbidity and mortality rates due to colorectal cancer (CRC) compared to White Americans. While the causes of these disparities are complex, regular screening can help reduce them. However, adherence to CRC screening guidelines remains low, particularly among African Americans.

One strategy to reduce CRC screening disparities is using strategic communication interventions to promote the fecal immunochemical test (FIT). FIT is a low-cost, non-invasive screening method that alleviates common patient barriers to CRC screening and is as effective as colonoscopy in reducing CRC incidence and mortality.

Tailored messaging interventions have been shown to improve CRC screening rates. However, two critical questions must be addressed before implementing tailored screening interventions within healthcare systems: (1) To what extent must message content be tailored to be effective? and (2) How can participants be effectively engaged?

This study builds upon an existing project that utilizes mobile Virtual Human Technology (VHT) to deliver tailored CRC screening messages. Virtual Human Agents (VHAs) provide a unique opportunity to customize communication strategies, including linguistic adaptation, to align with patient preferences. Such interventions can help mitigate CRC screening barriers such as cultural mismatch and low self-efficacy.

This study investigates explicitly the role of dialectal linguistic features in shaping willingness to be screened for CRC. The pilot study is exploratory in nature and seeks to examine the following aim: To assess how tailoring the dialectal variety of VHA speech affects willingness to be screened for CRC.

We aim to recruit 750 participants, each of whom will interact with a VHA that varies in speech style across four conditions: (1) non-dialectal linguistic features, (2) a low-level integration of dialectal linguistic features, (3) a high-level integration of dialectal linguistic features, or (4) a voiceless, text-only control. Following the interaction, participants will assess the VHA's credibility using survey-based measures.

ELIGIBILITY:
Inclusion Criteria:

* Out of guidelines for colorectal cancer screening
* No fecal immunochemical test within the last 12 months
* No colonoscopy within the last ten years)

Exclusion Criteria:

* Must meet inclusion criteria

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Krieger, PhD, Principal Investigator — Mayo Clinic of Jacksonville; Kevin Tang, PhD, Principal Investigator — University of Florida
Locations (1):
- Qualtrics, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Text-only: A virtual health assistant that will consist of photos of the computer-generated doctor with text that will guide participants through the interaction. No voice will accompany the photos or text.
  Text-only: virtual health assistant that will consist of photos of the computer-generated doctor with text that will guide participants through the interaction. No voice will accompany the photos or text.
Period: Overall Study
Arm/Group | Text-only | High Dialectal | Low Dialectal | Non-Dialectal
Started | 107 | 214 | 212 | 218
Completed | 107 | 214 | 212 | 218
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text-only | High Dialectal | Low Dialectal | Non-Dialectal | Total
Number analyzed (Participants) | 107 | 214 | 212 | 218 | 751
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 176 | 158 | 168 | 577
  >=65 years | 32 | 38 | 54 | 50 | 174
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 104 | 108 | 110 | 376
  Male | 53 | 110 | 104 | 108 | 375
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 107 | 214 | 212 | 218 | 751
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 107 | 214 | 212 | 218 | 751

OUTCOME MEASURES:

1. Primary Outcome: Intention to Talk to Doctor About Colorectal Cancer Screening
Description: Measure: Intention to talk to a doctor about colorectal cancer screening. Construct: Behavioral intention to communicate Item: The virtual appointment made me want to discuss colon cancer screening options with my doctor.
  Participants will respond using three 5-point Likert scales that will be summed. The total score ranges from 3 to 15, with higher scores indicating a greater intention to discuss colorectal cancer screening with a healthcare professional. Mean scores closer to 3 reflect lower intention, while mean scores closer to 15 reflect higher intention.
Time Frame: Immediately after the intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Text-only | High Dialectal | Low Dialectal | Non-Dialectal
Number analyzed (Participants) | 107 | 214 | 212 | 218
units on a scale | 11.42 (3.43) | 11.31 (3.55) | 11.87 (3.27) | 11.42 (3.38)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 weeks.
Description: During the study, 751 participants were monitored/assessed for other (non-serious) adverse events, but none were observed.
Arm/Group | Text-only | High Dialectal | Low Dialectal | Non-Dialectal
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/214 | 0/212 | 0/218
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/214 | 0/212 | 0/218
Other Adverse Events (participants affected / at risk) | 0/107 | 0/214 | 0/212 | 0/218

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT04705363/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT04705363/ICF_001.pdf